CLINICAL TRIAL: NCT00084058
Title: A Phase I/II Safety, Tolerability, and Pharmacokinetic Study of High Dose Lopinavir/Ritonavir With or Without Saquinavir in HIV-Infected Pediatric Subjects Previously Treated With Protease Inhibitors
Brief Title: Safety of Saquinavir and High Doses of Lopinavir/Ritonavir in Children With HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1038; 10045 (Registry Identifier: DAIDS ES); PACTG P1038
Record Dates: First submitted 2004-06-04; First posted 2004-06-07 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose Intensification; Pharmacokinetic Sampling; Treatment Experienced; Child
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Saquinavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Saquinavir

SUMMARY:
The purpose of this study is to determine the effect of increased doses of lopinavir/ritonavir (LPV/r) and saquinavir (SQV) in HIV infected children who are failing their current antiretroviral regimen

DETAILED DESCRIPTION:
Since current drugs cannot cure HIV infection, lifelong therapy is required. Development of drug resistance is common, with 30% to 80% of patients with initial viral load decreases following a potent anti-HIV regimen experiencing regimen failure within the first year of therapy. Dose intensification (increasing dosing of treatment medications) has been used successfully in pediatric oncology. Dose intensification in HIV infected patients may overcome resistance and, as similarly observed in cancer, may result in a greater rate of viral inhibition, maximizing the degree and durability of viral suppression. This study will evaluate dose intensification in HIV infected children and adolescents who are failing their current antiretroviral regimen and have significant genotypic and phenotypic resistance.

Participants in this 3-step study will have previously undergone genotypic resistance testing as part of their regular clinical care. Participants will have phenotypic resistance testing done at screening or within 6 months prior to study entry. Participants in this study will have either a genotypic profile with at least 4 of the required protease mutations or phenotypic resistance to LPV that is at least fivefold greater than wild type while on a failing regimen within 6 months of study screening.

In Step 1, Group 1 participants will be randomly assigned to either a drug regimen without a nonnucleoside reverse transcriptase inhibitor (NNRTI) or a drug regimen with an NNRTI for Group 2 participants. Participants and their doctors will work with study investigators to select the best treatment regimen possible. All participants in the study will receive LPV/r as part of their drug regimens. Participants in Group 1 will take a higher dose of LPV/r than participants in Group 2 because NNRTIs lower LPV/r levels in the blood.

At Week 2, participants will undergo a 12-hour pharmacokinetic (PK) test to evaluate the drug levels in their blood. If LPV/r levels are not high enough to control HIV and the participant can swallow tablets, hard gel capsules, or the contents of hard gel capsules with food or milk, the participant will begin taking SQV as part of his or her drug regimen and enter Step 2. After two weeks of taking SQV, participants will again undergo PK testing at Week 6. Based on these test results, the dose of SQV will then be increased, decreased, or maintained. Participants who do not add SQV to their regimen will continue taking LPV/r for the remainder of the study and stay in Step 1. If the PK test indicates SQV blood concentrations are sufficient, the participant will remain in Step 2. If the PK test indicates SQV blood concentrations are too low, the SQV dose will be increased and the participant will enter Step 3. After 2 weeks of taking elevated doses of SQV, participants will undergo PK testing at Week 10. If the PK test indicates that SQV blood concentrations are too high, the SQV dose will be decreased. At Week 14, participants who receive a reduced SQV dose will again undergo PK testing to verify that SQV blood concentrations are optimal.

Participants will have study visits at Weeks 2, 4, 6, 7, and 8, then every 4 weeks through the end of the study at Week 48. Study visits will include a physical exam, health history assessment, and blood collection. Blood collection for PK studies will occur at selected visits. Study visits at Weeks 2 and 12 will include an electrocardiogram (ECG or EKG).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* HIV RNA viral load greater than 5,000 copies/ml
* At least 6 months of continuous therapy with a protease inhibitor (PI) prior to study entry
* No change in antiretroviral therapy since genotypic resistance testing
* Genotypic resistance testing indicating a primary protease mutation at position 32, 47, 48, 50, 82, or 84 and at least three other mutations in positions 10, 20, 24, 30, 32, 33, 36, 46, 47, 48, 50, 53, 54, 71, 73, 77, 82, 84, or 90 OR phenotypic resistance testing, within 6 months of screening while on a failing regimen, indicating at least a fivefold increase in LPV as compared to wild type HIV
* Parent or legal guardian willing to provide informed consent
* If sexually active, agree to use acceptable methods of contraception
* Have a telephone, pager, or other method of reliable communication with study staff
* Able and willing to swallow study medications

Exclusion Criteria:

* Any drug toxicity greater than Grade 3 at screening
* Certain abnormal laboratory values
* Acute opportunistic or serious bacterial infection requiring treatment
* Chemotherapy for active cancer
* Any significant diseases (other than HIV infection) that may, in the opinion of the investigator, interfere with the study
* Require certain medications
* History of heart problems
* Family history of prolonged QTc-Interval Syndrome or prolonged QTc-interval at study entry
* Pregnancy or breastfeeding

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Life-threatening adverse events attributable to study drugs
dose-limiting toxicity, defined as adverse events of Grade 3 or greater attributable to study drug and require dose reduction or interruption but are not judged to be life-threatening by the protocol team

SECONDARY OUTCOMES:
Pharmacological success, defined as achieving an inhibitory quotient (IQ) of 15 after 2 weeks on high-dose LPV/r without life-threatening or dose-limiting toxicity
virologic success, defined by optimal response (undetectable viral load) at Week 24 or adequate response (0.75 log drop in viral load or more) from baseline to Week 24
immunologic success, defined as a CD4% increase from baseline of 5% or more points by Week 24
minimal criterion for overall success, defined as a 0.75 log drop in viral load or more or 5% point increase in CD4% from baseline to Week 24
virologic failure, defined as an inadequate (less than 0.75 log drop in viral load) or suboptimal (confirmed viral load of greater than 400 copies/ml) response at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Havens, MD, Study Chair — Medical College of Wisconsin
Locations (15):
- United States (13):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Foster C, Lyall EG. Children with HIV: improved mortality and morbidity with combination antiretroviral therapy. Curr Opin Infect Dis. 2005 Jun;18(3):253-9. doi: 10.1097/01.qco.0000168387.24142.cf. PMID 15864104
- [Background] Havlir DV, Gilbert PB, Bennett K, Collier AC, Hirsch MS, Tebas P, Adams EM, Wheat LJ, Goodwin D, Schnittman S, Holohan MK, Richman DD; ACTG 5025 Study Group. Effects of treatment intensification with hydroxyurea in HIV-infected patients with virologic suppression. AIDS. 2001 Jul 27;15(11):1379-88. doi: 10.1097/00002030-200107270-00007. PMID 11504959
- [Background] Kempf DJ, Isaacson JD, King MS, Brun SC, Sylte J, Richards B, Bernstein B, Rode R, Sun E. Analysis of the virological response with respect to baseline viral phenotype and genotype in protease inhibitor-experienced HIV-1-infected patients receiving lopinavir/ritonavir therapy. Antivir Ther. 2002 Sep;7(3):165-74. PMID 12487383
- [Background] Kulkosky J, Nunnari G, Otero M, Calarota S, Dornadula G, Zhang H, Malin A, Sullivan J, Xu Y, DeSimone J, Babinchak T, Stern J, Cavert W, Haase A, Pomerantz RJ. Intensification and stimulation therapy for human immunodeficiency virus type 1 reservoirs in infected persons receiving virally suppressive highly active antiretroviral therapy. J Infect Dis. 2002 Nov 15;186(10):1403-11. doi: 10.1086/344357. Epub 2002 Oct 29. PMID 12404155
- [Result] Malee K, Williams PL, Montepiedra G, Nichols S, Sirois PA, Storm D, Farley J, Kammerer B; PACTG 219C Team. The role of cognitive functioning in medication adherence of children and adolescents with HIV infection. J Pediatr Psychol. 2009 Mar;34(2):164-75. doi: 10.1093/jpepsy/jsn068. Epub 2008 Jul 22. PMID 18647794
- [Result] Robbins BL, Capparelli EV, Chadwick EG, Yogev R, Serchuck L, Worrell C, Smith ME, Alvero C, Fenton T, Heckman B, Pelton SI, Aldrovandi G, Borkowsky W, Rodman J, Havens PL; PACTG 1038 Team. Pharmacokinetics of high-dose lopinavir-ritonavir with and without saquinavir or nonnucleoside reverse transcriptase inhibitors in human immunodeficiency virus-infected pediatric and adolescent patients previously treated with protease inhibitors. Antimicrob Agents Chemother. 2008 Sep;52(9):3276-83. doi: 10.1128/AAC.00224-08. Epub 2008 Jul 14. PMID 18625762